CLINICAL TRIAL: NCT00005880
Title: A Phase II Trial of Inhaled Budesonide (Pulmicort Turbuhaler) in Persons With Dysplasia of the Bronchial Epithelium
Brief Title: Budesonide in Treating Former and Current Smokers With Bronchial Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000067919; BCCA-CIC-98-37; UBC-C98-0411; NCI-P00-0147
Record Dates: First submitted 2000-06-02; First posted 2004-02-25 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-07

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Budesonide

INTERVENTIONS:
Drug: budesonide

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of budesonide may be an effective way to prevent bronchial dysplasia.

PURPOSE: Randomized double-blinded phase II trial to determine the effectiveness of budesonide in treating former or current smokers who have bronchial dysplasia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of inhaled budesonide on the number and grade of bronchial epithelial dysplastic lesions in former and current smokers. II. Compare the effect of inhaled budesonide vs placebo in modulating several intermediate biomarkers (i.e., proliferation, apoptosis, morphometric, and methylation markers) in this patient population. III. Correlate the regression of bronchial dysplasia (number and grade) and improvement in sputum cytology (morphometric grade of atypical cells) with the modulations in molecular biomarkers in this patient population. IV. Compare the stability of the chemopreventive effect of these treatment regimens at six months after completion of these regimens in these patients. V. Compare the safety of these treatment regimens in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are stratified according to gender, smoking status (current vs former), and morphometric index (no greater than 3.4 vs greater than 3.4). Patients are randomized into one of two treatment arms. Arm I: Patients receive inhaled budesonide twice daily. Arm II: Patients receive an inhaled placebo twice daily. Treatment continues for 6 months in the absence of disease progression or unacceptable toxicity. Patients are followed at 7 months and 12 months.

PROJECTED ACCRUAL: A total of 110 patients (55 per treatment arm) will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed mild, moderate, or severe bronchial dysplasia More than one suspicious area of abnormal fluorescence on bronchoscopy If only one abnormal area, lesion must be greater than 1.5 mm Current or ex-smokers who have smoked at least 30 pack years (e.g., 1 pack per day for at least 30 years) Sputum cells with morphometric index at least 7 by computer-assisted image analysis No invasive cancer on bronchoscopy or abnormal chest x-ray suspicious of lung cancer

PATIENT CHARACTERISTICS: Age: 40 to 74 Performance status: Not specified Life expectancy: Not specified Hematopoietic: No bleeding disorder Hepatic: Not specified Renal: Not specified Cardiovascular: No unstable angina or congestive heart failure Pulmonary: No active pulmonary tuberculosis No acute bronchitis or pneumonia No acute or chronic respiratory failure Other: No history of allergy to budesonide or lactose No known reaction to lidocaine Ability to reliably take medication Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: At least 6 months since prior oral glucocorticoids (e.g., prednisone) At least 6 months since prior inhaled glucocorticoids (e.g., budesonide, Beclovent, or Becloforte) Radiotherapy: Not specified Surgery: Not specified

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Study Chair — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada